CLINICAL TRIAL: NCT01690169
Title: Investigation on Safety, Tolerability, and Pharmacokinetics of Single Doses of NNC0113-0987 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9927-3909; 2012-000047-27 (EudraCT Number); U1111-1126-7584 (Other: WHO)
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0113-0987 (Experimental)
  Interventions: Drug: NNC0113-0987
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0113-0987 — A single dose for oral administration, up to 7 dose levels will be investigated. If a non-tolerated dose level has been reached, the dose level will not be increased further.
  Arms: NNC0113-0987
Drug: placebo — A single dose of oral placebo administered.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) of single doses of NNC0113-0987 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with good general health as judged by the investigator, based on medical history, physical examination including 12-lead electrocardiogram (ECG), vital signs, and blood assessments at the screening visit
* Body mass index (BMI) above or equal to 18.5 and below 30 kg/m^ 2

Exclusion Criteria:

* Male subjects who are sexually active and not surgically sterilised, who or whose partner is unwilling to use two different forms of effective contraception, one of which has to be a barrier method (e.g., condom with spermicidal foam/gel/film/cream) for the duration of the trial and for 12 weeks following the last dose of trial medication
* Participation in another trial within 90 days prior to screening
* Subjects with a history of or presence of cancer, diabetes, or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal (including gastroesophageal reflux disease and irritable bowel syndrome), endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorders that might have an impact on the current trial, as judged by the investigator
* Subjects who are known to have hepatitis or who are carriers of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies, or have a positive result to the test for Human Immunodeficiency Virus (HIV) antibodies
* History of acute idiopathic or chronic pancreatitis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09-14 (Actual); Primary Completion 2012-12-11 (Actual); Study Completion 2012-12-11 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From the dosing visit and until completion of the post-treatment follow-up visit (i.e. day 12-25)

SECONDARY OUTCOMES:
Number and severity of hypoglycaemic episodes | From dosing visit and until completion of the post-treatment follow-up visit (i.e. day 12-25)
AUC, the area under the NNC0113-0987 plasma concentration-time curve | From dosing visit to infinity
Cmax, the maximum plasma concentration of NNC0113-0987 | From dosing visit until last PK sampling visit (e.g. day 11)
tmax, the time to maximum plasma concentration of NNC0113-0987 | From dosing visit until last PK sampling visit (e.g. day 11)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Nottingham, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com